CLINICAL TRIAL: NCT04141306
Title: Radioiodine-avid Bone Metastases From Differentiated Thyroid Cancer Without Structural Abnormality, a Singular Entity With Heterogeneous Outcomes.
Brief Title: Radioiodine-avid Bone Metastases From Thyroid Cancer Without Structural Abnormality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_1919
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Bone Metastases; Thyroid Cancer
Keywords: Radioiodine Bone Metastases; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Administrative data — Evaluation of month and year of birth, sex, referent doctor and surgeon
Other: Clinical data — Evaluation of diagnostic circumstances, vital status at last follow up
Other: Histological data — Evaluation of Pathology report of thyroid surgery
Other: Imaging data — Evaluation of scintigraphy, MRI, scan
Other: Biological data — Evaluation of thyroglobulin, antithyroglobulin antibodies
Other: Further treatment — Evaluation of surgery, radiotherapy, targeted therapy

SUMMARY:
Bone radioiodine (RAI) uptake without structural abnormality in thyroid cancer (TC) patients may be related to false positive or to microscopic foci of metastatic tissue. In such cases, outcome is reported to be excellent.

Indeed, Robenshtok et al. reported a serie of patients with RAI-avid bone metastases of TC without structural abnormality on imaging studies who have more favorable long-term prognosis than those harbouring structurally visible bone metastases and do not undergo skeletal-related complications.

The investigators report the case of Mrs D., who had been operated for a pathologic tumor stage 3: pT3(m) poorly differentiated TC at the age of 43. The first post-therapeutic whole body scan revealed 3 foci of bone uptake (right clavicle, L2, L3). The elevated level of thyroglobulin (157ng/mL) favoured the hypothesis of bone metastases despite the absence of any structural lesion on CT and MRI. She received 7 courses of radioiodine therapy. The right clavicle RAI uptake persisted, and subsequent CT disclosed an osteolytic lesion which was treated by radiofrequency and external beam radiation. Twenty-five years after the diagnosis, she has a persistent morphological disease with a 30x8mm progressive lesion on the right clavicle, for which surgery is planned.

The aim of the present study is to describe the natural history and evolution of radioiodine avid bone metastases from thyroid cancer without structural abnormalities and to identify prognosis factors.

ELIGIBILITY:
Inclusion Criteria:

* Differentiated thyroid cancer
* Ablation therapy with post dose scintigraphy
* At least one radioiodine bone uptake without structural correlation on high-resolution imaging

Exclusion Criteria:

* A single radio iodine bone uptake with structural correlation on imaging
* Diagnosis of bone metastasis after a skeletal related event including spinal cord compression, pathological fracture, need for external beam radiation, surgery to bone, or development of hypercalcemia of malignancy
* Follow up less than 6 months
* Missing data in medical record

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received total thyroidectomy in a context of differentiated thyroid cancer showing at post-therapy scintigraphy at least one radioiodine bone uptake without structural correlation on high-resolution imaging
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission of thyroid cancer | 1 month
  * Disappearance of pathologic radio iodine uptake, including bone uptake, on post-therapy scintigraphy
  * No structural evidence of disease on high-resolution imaging
  * Suppressed serum Tg < 0.6 ng/mL, no detectable TgAb (thyroglobulin antibody)